CLINICAL TRIAL: NCT03909204
Title: Laparoscopic-Assisted Percutaneous Endoscopic Cecostomy (LAPEC) in Adults for the Treatment of Severe Constipation
Brief Title: LAPEC for the Treatment of Severe Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Trnava (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAPEC for obstipation
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Cecostomy; Complications; Constipation
Keywords: Laparoscopic-Assisted Percutaneous Endoscopic Cecostomy
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Masking Description: Supportive Care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LAPEC (Other): Patients with cecal percutaneous catheter placement.
  Interventions: Procedure: LAPEC

INTERVENTIONS:
Procedure: LAPEC — Laparoscopic-Assisted Percutaneous Endoscopic Cecostomy: Initially, one to tree-laparoscopy port technique will be used, with hand placement of seroperitoneal sutures for cecal fixation. After than during colonoscopy a cecal position will be visualized and colonic lumen will be insuflated. After than the PEC tube will be introduced into the cecum using the dilators and sheath. Intravenous antibiotics will be given prior to the procedure and will continued parental temporary and later orally after catheter insertion. One weeks later, antegrade colonic enema will start during an out-patient visit including an educational training of the patient to the catheter manipulation. Antegrade enema solution will start at dose of 2ml/kg and will be increased up to 20ml/kg or a maximum dose of 2000 mL daily. Adjuvant of colonic motility stimulants are allowed during follow-up.
  Other Names: Laparoscopic-Assisted Percutaneous Endoscopic Cecostomy

SUMMARY:
Effective treatment for constipation is a real clinical challenge especially in patients with severe symptoms. Dietary measures (bulking agents) and drugs (laxatives, stool softeners, suppositories and enemas etc.) have limited efficacy in severe cases. If conservative measures do not help, surgical therapies might be considered. Subsequently, antegrade enemas through percutaneous colonic catheter were introduced as a less invasive option for treating severe constipation. The cecostomy has been performed laparoscopically, percutaneously, and with the laparoscopic-assisted percutaneous endoscopic cecostomy (LAPEC) technique. This approach allows patients to deliver osmotic agents to the right colon.The procedure has been demonstrated to be safe and effective in young adults and pediatrics. To date, there are only few studies evaluating the safety and efficacy of the LAPEC procedure in adults and all have retrospective profile. The aim of this prospective study is to compare short and long-term efficacy and safety of LAPEC in patients with severe constipation. Symptoms of defecation will be the main outcome criteria.

ELIGIBILITY:
Inclusion Criteria:

* Refractory (> 6 months) and severe (based on a =KESS >11) and non-invasive therapeutic approaches, including an enhanced fiber diet, lifestyle changes, laxatives, and biofeedback failed.
* Slow transit constipation
* Anorectal malformation
* Mixed constipation (combination of outlet obstruction and slow transit)
* Hirschsprung's disease
* Idiopathic constipation ineffective to standard treatment
* Cauda equine syndrome
* Combination of spina bifida and tethered cord
* Colonic neuropathy.
* Persons 18 years or older at the time of signing the informed consent
* Signed informed consent

Exclusion Criteria:

* Non-LAPEC cecostomy procedure
* Pre-existing severe electrolyte imbalance
* Chronic high rectal tone
* Advanced liver cirrhosis (Child B or Child C)
* Pregnancy or puerperium
* Advanced colorectal cancer
* Presence of ventriculoperitoneal shunt
* Colonic disease or surgery that might impact safety of percutaneous colostomy tube placement (right hemicolectomy, IC resection, previous apendicostomy) and confirmed inflammatory bowel disease
* Any other condition, which in the opinion of the investigator would interfere with study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Change in Bowel QoL | Exit data will be collected at 3 and 6 months after Intake data collection / PEC placement
  Main outcome is the proportion of patients with treatment success at 3 and 6 months after the catheter placement. Treatment success is defined as a decrease of Quality of Life symptoms score at least 50% to a baseline values. To assess constipation severity the Knowles Eccersley Scott Symptom (KESS) before and throughout the study will be completed. The KESS is an 11-item tool for diagnosis of constipation. The KESS uses four- to five-point Likert scales that are scored on an unweighted linear integer scale. Total scores can range from 0 (no symptoms) to 39 (high symptom severity).

SECONDARY OUTCOMES:
Change in Bowel QoL | 3 months, 6 months, 12 months, 24 months
  Evolution of Quality of Life questionnaire before and after PEC placement at 3, 6, 12 and 24 months. To assess constipation severity the Knowles Eccersley Scott Symptom (KESS) before and throughout the study will be completed. The KESS is an 11-item tool for diagnosis of constipation. The KESS uses four- to five-point Likert scales that are scored on an unweighted linear integer scale. Total scores can range from 0 (no symptoms) to 39 (high symptom severity).
Removal rate | 12 months
  Proportion of patients with PEC in use and removed.
Transit time | At 3 and 12 month after PEC placement
  Change in x-ray transit time
Frequency and Severity of Abdominal Pain | Data collection will start following consent and procedural training and will be collected daily from day 1 for the duration of the study, an expected average of 12 weeks
  Frequency and severity of abdominal pain will be recorded daily and measured using the Visual analog pain scale as the appropriate visual analog scale. Score is based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-points line that represents a continuum between the two ends of the scale-"no pain" on the left end (0) of the scale and the "worst pain" on the right end of the scale (10).
Flush Administration Time | Data collection will start with the first flush administered following discharge from the hospital and will be collected with every subsequent flush through completion of the study, an expected average of 48 weeks
  Administration time in minutes per flush will be defined as the time at which the tubing connected to the bag or syringe and the cecostomy fluid starts to infuse into the patient to the time the infusion is completed.
Flush volume | Data collection will start with the first flush administered following discharge from the hospital and will be collected with every subsequent flush through completion of the study, an expected average of 48 weeks
  Volume will be measured and recorded by the patient with each flush and calculated by the investigator in mL/kg using the weight obtained at the clinic visit preceding each effectiveness phase change.
Procedural adverse event | 1 month
  Perioperative adverse events (complications)
Long-term adverse events | 3, 6, 12, 24 months
  Incidence rate of adverse events during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Skuta, Principal Investigator — Surgeon
Locations (1):
- Rastislav Hustak, Trnava, Slovakia